CLINICAL TRIAL: NCT04149431
Title: Multicenter Double Blinded Placebo-controlled Randomized Study to Evaluate Clinical Efficacy, Tolerability, Safety of Medical Product Derinat®, Solution for External and Local Use 0.25% in Acute Infections of Respiratory System in Children
Brief Title: Multicenter Study to Evaluate Efficacy, Tolerability, Safety of Derinat
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PharmPak, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ДК-18
Record Dates: First submitted 2019-10-16; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Respiratory Infections in Children
Keywords: Derinat; Respiratory infection; Children
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Derinat

STUDY DESIGN:
Intervention Model Description: This is a multi-center, double-blind, randomized phase III-IV clinical trial in parallel groups to evaluate the efficacy and safety of Derinat versus Placebo in patients with acute upper respiratory tract infection.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind randomized placebo controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Derinat (Active Comparator): nasal drops
  Interventions: Drug: Derinat
- Placebo (Placebo Comparator): nasal drops
  Interventions: Drug: Derinat

INTERVENTIONS:
Drug: Derinat — desoxyribonucleate sodium
  Other Names: desoxyribonucleate sodium

SUMMARY:
This multicenter prospective double blinded placebo-controlled randomized study is designed to to evaluate clinical efficacy, tolerability and safety of medical product Derinat®, solution for external and local use 0.25% in acute infections of respiratory system in children

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized phase III-IV clinical trial in parallel groups to evaluate the efficacy and safety of Derinat versus Placebo in patients with acute upper respiratory tract infection.

The study will include only patients with mild to moderate acute upper respiratory tract infection, without complications. According to the recommendations of the FDA (Guidance for Industry Influenza: Developing Drugs for Treatment and/or Prophylaxis) this category of patients is the best suited for placebo-controlled studies, because the expected serious risks without treatment are negligible. For studies evaluating the therapy of patients with mild to moderate acute respiratory upper respiratory tract infection without complications, a placebo-controlled trial design is preferred, as opposed to designs with no less efficacy (non-inferiority).

This study provides for the inclusion of both outpatient patients and patients admitted to the hospital for epidemiological indications (i.e. patients with acute respiratory infection of the upper respiratory tract of mild and moderate severity without complications that pose an epidemic risk.

Assessment of criteria of severity of acute respiratory infection of the upper respiratory tract will be carried out by Investigator based on standards of diagnosis and treatment of infectious diseases in children at the stages of medical care, depending on the forms of severity of the disease.

The study is planned sequentially in 5 age groups. The study begins with the older age group and as the results on the safety of the drug are obtained, in the course of the study, it is possible to move to younger age groups

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Male and female patients.
3. The age of the child at the time of first intranasal administration of drug for age group 1: 12 years to <18 years; for age group 2: from 6 years to <12 years; for age group 3: from 2 years to <6 years; for age group 4: 7 months to <2 years; for age group 5: from 0 months to 6 months.
4. Outpatient and inpatient patients hospitalized for epidemiological reasons, with a diagnosis of acute respiratory infection of the upper respiratory tract of mild to moderate severity. (ICD 10: J00 - J06 Acute respiratory infections of the upper respiratory tract).
5. The positive result of the enzyme immunoassay express test for pathogens of acute respiratory infection of the upper respiratory tract on screening.
6. At least one episode of body temperature up to 38C and above within 48 hours prior to screening.
7. Presence of at least one of the following mild to moderate symptoms at screening: headache, weakness/malaise, muscle pain/aching, feeling of heat/chills.
8. The duration of the disease is not more than 48 hours at the time of screening according to the patient/parents/adoptive parents.
9. Adequate contraceptive methods during the study for the patients with childbearing potential

Exclusion Criteria:

1. Positive express test (in urine) for pregnancy in patients with childbearing potential (menarche).
2. Individual intolerance or hypersensitivity to any of the components of the drug according to the medical history.
3. Taking any drugs with immunomodulatory effect less than 30 days before screening according to medical history.
4. The presence of complications of acute respiratory infection of the upper respiratory tract, signs of severe disease at the time of screening (fever more than 39ºC, febrile convulsions).
5. Acute infectious diseases: diphtheria, measles, infectious mononucleosis, herpes type 1 and 2, rubella, scarlet fever, acute BGSA-tonsillopharyngitis at the time of screening or 30 days before screening.
6. Chronic diseases of the respiratory system (Bronchial asthma, COPD).
7. HIV infection, chronic viral hepatitis B or C (according to history).
8. Impaired renal function with serum creatinine level more than 1.5 times higher than the upper limit of the normal range.
9. Severe liver failure or active liver disease (including viral hepatitis B or C) and increase of ALT and AST more than 5 times of upper limit of the normal range.
10. Participation in any clinical trials and / or taking an experimental drug within 30 days prior to the screening visit.
11. Other significant diseases and conditions of the patient, including mental and physical diseases

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 350 (Estimated)
Dates: Start 2019-12-15 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Superiority of Derinat | through study completion, an average of 30 days
  Assessment of frequency of resolution of symptoms of acute respiratory infection of the upper respiratory tract confirmed by the absence of symptoms (0 points on the scale of evaluation of symptoms of acute upper respiratory infection during at least 24 hours

SECONDARY OUTCOMES:
Efficacy of Derinat | through study completion, an average of 30 days
  Assessment of frequency of resolution of symptoms of acute upper respiratory infection? time from start of investigational therapy to resolution of symptoms of acute upper respiratory infection and assessment of frequency of elimination of pathogens of acute respiratory infections of the upper respiratory tract from the mucous membrane of the nasopharynx and oropharynx to Day 8
Safety of Derinat | through study completion, an average of 30 days
  Assessment of incidence of complications in acute upper respiratory tract infection and the incidence of adverse events and serious adverse events of varying severity according to subjective complaints, laboratory tests, physical examination, assessment of vital signs and electrocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Irina Gerasimova, Dr., Study Director — PharmPak, LLC
Locations (1):
- Irina Gerasimova, Moscow, Russia